CLINICAL TRIAL: NCT05796128
Title: Nasal Intermittent Positive Pressure Ventilation Versus Nasal Continuous Positive Airway Pressure Durante la Somministrazione Del Surfattante Con Tecnica LISA
Brief Title: NIPPV vs.nCPAP During LISA Procedure
Acronym: NIPAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Carlo Dani, Full Professor of Pediatrics, University of Florence
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIPAL02
Record Dates: First submitted 2023-03-08; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Respiratory Distress Syndrome, Newborn
Keywords: Surfactant; LISA procedure; Preterm infant
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Premature Birth | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LISA with NCPAP (Active Comparator): In this group, infants will receive NCPAP during LISA procedure.
  Interventions: Procedure: Nasal continuous positive airway pressure (NCPAP)
- LISA with NIPPV (Experimental): In this group, infants will receive NIPPV during LISA procedure.
  Interventions: Procedure: Nasal Intermittent Positive Pressure Ventilation (NIPPV)

INTERVENTIONS:
Procedure: Nasal Intermittent Positive Pressure Ventilation (NIPPV) — In this group, infants will receive NIPPV during LISA procedure.
  Arms: LISA with NIPPV
Procedure: Nasal continuous positive airway pressure (NCPAP) — In this group, infants will receive NCPAP during LISA procedure.
  Arms: LISA with NCPAP

SUMMARY:
The goal of this randomized controlled study is to compare the efficacy of using NIPPV versus NCPAP during the LISA procedure in very preterm infants.

The main question it aims to answer is:

• Does NIPPV during the LISA procedure decrease the need for a second dose of surfactant or the need of mechanical ventilation during the first 72 hours of life in comparison with NCPAP? Infants with gestational age between 25+0 and 31+6 weeks of gestation with RDS who do not require VM and treated with NCPAP and FiO2 >0.30 within the first 6 hours of life who received the first dose of caffeine will be eligible for enrollment in the study Participants will be randomized to receive surfactant with conventional LISA procedure, i.e. performed during NCPAP, or with LISA procedure performed during NIPPV.

ELIGIBILITY:
Inclusion Criteria:

* -Infants with gestational age between 25+0 and 31+6 gestational weeks,
* -RDS which does not require MV
* -Treatment with NCPAP and FiO2 >0.30 within the first 6 hours of life,
* -First dose of caffeine administered

Exclusion Criteria:

* -absence of informed consent,
* -major congenital malformations,
* -hydrops fetalis,
* -chromosomal diseases,
* -previous treatment with surfactant,
* -cardiorespiratory instability requiring treatment with vasoactive drugs,
* -pneumothorax,
* -death within 72 hours of life.

Ages: 0 Hours to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 202 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-01-23 (Actual)

PRIMARY OUTCOMES:
Surfactant or mechanical ventilation | The need for a second dose of surfactant or mechanical ventilation will be evaluated within the first 72 hour of life
  Need for a second dose of surfactant or mechanical ventilation

SECONDARY OUTCOMES:
Noninvasive ventilation | Participants will be monitored for the duration of their hospital stay, which is an average of 10 weeks
  Duration of noninvasive ventilation
Mechanical ventilation | Participants will be monitored for the duration of their hospital stay, which is an average of 10 weeks
  Duration ofmechanical ventilation
Bronchopulmonary dysplasia | Participants will be monitored for the duration of their hospital stay, which is an average of 10 weeks
  Frequency of mild, moderate, and severe bronchopulmonary dysplasia

CONTACTS AND LOCATIONS:
Locations (1):
- Careggi University Hospital, Division of Neonatology, Florence, Italy

IPD SHARING:
Plan to Share IPD: Undecided